CLINICAL TRIAL: NCT00411190
Title: A Study to Evaluate the Potential for Pharmacokinetic Interaction Between SB 462795 and SSRIs in Healthy Subjects [3A]
Brief Title: Study To Determine The Effects Of Doses Of Relacatib On The Metabolism Of Acetaminophen, Ibuprofen And Atorvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SB-462795/008
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Postmenopausal; Osteoporosis
MeSH Terms: conditions — Osteoarthritis; Osteoporosis | interventions — relacatib; Acetaminophen; Ibuprofen; Atorvastatin

ARMS (2):
- Session 1 (Experimental): Subjects will receive 500 mg acetaminophen on Day 1, 400 mg ibuprofen on Day 2, 40 mg atorvastatin on Day 3.
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen; Drug: Atorvastatin
- Session 2 (Experimental): Subjects will be randomized to receive relacatib 60 mg or 120 mg from Day 1-14. On Day 15 subjects will receive 500 mg acetaminophen, 400 mg ibuprofen on Day 16 and 40 mg atorvastatin on Day 17 with usual dose of relacatib.
  Interventions: Drug: Relacatib; Drug: Acetaminophen; Drug: Ibuprofen; Drug: Atorvastatin

INTERVENTIONS:
Drug: Relacatib — Subjects will administer 60 or 120 mg tablets in Session 2
  Arms: Session 2
Drug: Acetaminophen — Acetaminophen will be administered orally
Drug: Ibuprofen — Ibuprofen will be administered orally
Drug: Atorvastatin — Atorvastatin will be administered orally

SUMMARY:
Relacatib is being developed for the treatment of osteoporosis, osteoarthritis and possibly other bone disorders. Recent results suggest that relacatib interacts with the way our bodies metabolise drugs and so some drugs which are commonly prescribed to the intended target patient population could be affected by giving relacatib at the same time. The purpose of this study is to evaluate the effect of repeat dose administration of relacatib on the way subjects bodies metabolise three commonly prescribed medications in the osteoarthritis population: ibuprofen, acetaminophen, and atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Postmenopausal
* Body weight > 50 kg
* Body mass index (BMI) between 19 and 30
* The subject is willing and able to give a signed and dated written informed consent prior to admission to the study
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* Subjects with known morphea or sclerodermia
* Subjects with a history of myocardial infarction.
* Subjects with a history of renal/or hepatic disease unless the disease has been successfully treated and is no longer active; subjects with any evidence of renal/ or hepatic impairment on the screening physical and laboratory examination.
* Subjects with history of hypertension or systolic blood pressure
* Subjects with history of diabetes
* History of regular alcohol consumption exceeding 7 drinks/week (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
* History of use of tobacco- or nicotine-containing products within 6 months of screening, or a positive urine cotinine indicative of smoking at screening.
* Positive urine drug screen including alcohol (or alcohol breath test) at screening.
* Positive for HIV, hepatitis B virus or hepatitis C virus.
* Donation of blood in excess of 500 mL within 56 days prior to dosing
* History of sensitivity or contraindications to any of the study medications (i.e., relacatib, paracetamol, ibuprofen or atorvastatin) or components thereof.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Subjects whom are judged by the investigator to be at risk for acute angle closure glaucoma.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-10-19 (Actual); Primary Completion 2006-12-15 (Actual); Study Completion 2006-12-15 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to characterize the effect of relacatib at steady-state on the pharmacokinetics of a single oral dose of acetaminophen, ibuprofen and atorvastatin in healthy postmenopausal females. | Up to Day 17

SECONDARY OUTCOMES:
To assess the safety and tolerability of the concomitant administration of oral doses of relacatib and acetaminophen, ibuprofen and atorvastatin. To describe the changes from baseline in serum CTXI levels for each relacatib dose tested. | Up to Day 17

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Belgium (2):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Liège

REFERENCES:
- See also: Results for study SB-462795/008 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/SB-462795/008?search=study&search_terms=SB-462795%2F008#rs